CLINICAL TRIAL: NCT00983801
Title: A Phase II Study of Ixabepilone in Asian Subjects With Unresectable or Metastatic Gastric Cancer Previously Treated With Fluoropyrimidine-based Chemotherapy
Brief Title: Study of Ixabepilone in Asian Subjects With Unresectable or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-200
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixabepilone (Experimental)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Vial, Injection, Intravenous (IV), 40 mg/m^2, Every 21 days, Up to 8 cycles or until disease progression or intolerable toxicity. Additional treatment was given in agreement by both the investigator and sponsor. Ixabepilone 40 mg/m^2 was administered as a 3-hour IV infusion on Day 1 of each 21-day (3 week) cycle provided the participant met the retreatment criteria.
  Other Names: Ixempra; BMS-247550

SUMMARY:
The purpose of this study was to determine whether ixabepilone is effective in the treatment of unresectable or metastatic gastric cancer in Asian participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric carcinoma originating from the stomach or gastroesophageal junction
* Must have unresectable or metastatic disease
* Asian ethnicity
* Must have failed prior fluoropyrimidine-based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* measurable disease by with Response Evaluation Criteria in Solid Tumors (RECIST) guidelines

Exclusion Criteria:

* >1 prior chemotherapy regimen in the metastatic setting or >2 prior chemotherapy if subject also received adjuvant therapy
* Receipt of prior ixabepilone
* ECOG ≥2
* Known brain or meningeal metastasis
* Known viral hepatitis
* Prior taxane therapy
* Uncontrolled non-cancer related medical condition
* Second malignancy
* Peripheral neuropathy ≥ grade 2
* Inadequate hematologic, renal and hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- Local Institution, Hong Kong, Hong Kong
- Japan (2):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Sunto-Gun, Shizuoka
- Local Institution, Singapore, Singapore
- Local Institution, Seoul, South Korea
- Taiwan (2):
  - Local Institution, Taipei
  - Local Institution, Taoyuan Hsien

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 58 participants enrolled in this study, 6 failed screening criteria, and 52 received treatment.
Groups:
- Ixabepilone 40 mg/m^2 IV: ixabepilone 40 mg/m^2 intravenous (IV), every 21 days, up to 8 cycles or until disease progression or development of intolerable toxicity.
Period: Overall Study
Arm/Group | Ixabepilone 40 mg/m^2 IV
Started | 52 (Participants who received treatment.)
Completed | 52 (Participants who were taken off treatment.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
Age, Customized [Number; unit: participants]
  < 65 years | 40
  >=65 years | 12
  < 50 years | 9
  >=50 years | 43
Age, Customized [Median (Full Range); unit: years] | 56.5 [29.0 to 77.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 34
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 23
  Japanese | 15
  Korean | 13
  Asian Other | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — The ECOG PS is used to assess disease severity. A score of 0 is normal activity; 1=symptoms, but fully ambulatory; 2=symptomatic, but in bed <50% of the day; 3=needs to be in bed > 50% of the day, but not bedridden; 4=unable to get out of bed; 5=dead.
  participants
    0 (normal activity) | 20
    1 (symptoms, but fully ambulatory) | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR) Based on Modified Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) according to modified RECIST, as determined by investigator. CR: Disappearance of all evidence of target and non-target lesions. In case of lymph node, the lesions short axis of all nodes measuring <10 mm. PR: At least 30% reduction from baseline in the sum of the longest diameter (LD) of all target lesions. CR and PR criteria should be met again after 4 weeks and before 6 weeks after initial assessment. A 2-sided confidence interval (CI) was computed using Clopper-Pearson method.
Time Frame: During treatment, assessed every 6 weeks (± 1 week) starting from the 1st dose of therapy until disease progression, or development of intolerable toxicity, for a maximum of 8 cycles (maximum time that any participant was on therapy was 30 weeks)
Population: Response-evaluable participants: Participants who received at least 1 dose of ixabepilone with measurable disease at baseline and right cancer diagnosis (presence of histologic or cytologic diagnosis of advanced or metastatic adenocarcinoma originating in the stomach or gastroesophageal junction).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
percentage of participants | 15.4 [6.9 to 28.1]

2. Secondary Outcome: Time to Response
Description: Time to response is defined as the time in weeks from the first dose of study therapy until measurement criteria are first met for PR or CR (whichever status is recorded first). CR: Disappearance of all evidence of target and non-target lesions. In case of lymph node lesions, the short axis of all nodes should measure <10 mm. PR: At least 30% reduction from baseline in the sum of the LD of all target lesions. CR and PR criteria should be met again after 4 weeks and before 6 weeks of initial assessment.
Time Frame: Assessed every 6 weeks (± 1 week) starting from the first dose of study therapy until CR or PR (up to 12.1 weeks.)
Population: Participants who received at least 1 dose of study therapy and had a response of either CR or PR.
Measure: Median (Full Range); unit: weeks
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 8
weeks | 8.9 [5.1 to 12.1]

3. Secondary Outcome: Duration of Response
Description: Defined as the period in months from the time measurement criteria are first met for PR or CR until the first date of documented PD or death. Refer to outcome measure 1 for CR and PR. PD=≥20% increase in the sum of LD of target lesions and an absolute increase of at least 5 mm of tumor size in reference to the smallest sum LD recorded at or following baseline or the appearance of one or more new lesions or unequivocal progression of existing non-target lesions. Estimated by Kaplan-Meier product limit method and a 2-sided 95% CI for median duration was computed by Brookmeyer and Crowley method.
Time Frame: From the date of first PR or CR assessment to the date of progression, death, or last tumor assessment (maximum: 4.1 months)
Population: Participants who received at least 1 dose of ixabepilone and had either CR or PR. Participants who neither relapsed nor died were censored on the date of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 8
months | 3.1 [2.6 to 4.1]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS=the time interval from date of randomization to the earliest (first) progression or date of death. Participants who progressed or died were counted as events. PD=≥20% increase in sum of LD of target lesions and an absolute increase ≥5 mm in tumor size in reference to the smallest sum LD recorded at or following baseline or the appearance of one or more new lesions or unequivocal progression of existing non-target lesions. Estimated using the Kaplan-Meier product-limit method for all treated participants and a 2-sided 95% CI for the median PFS was computed by Brookmeyer and Crowley method).
Time Frame: From the date of initiation of study therapy to the date of progression (up to 8.1 months).
Population: Participants who received at least 1 dose of ixabepilone. Participants who died without reporting prior progression were considered to have progressed on their death day. Participants who did not progress or die were censored on their last tumor assessment day. Participants without on-study tumor assessments were censored at start date of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
months | 2.8 [2.1 to 3.5]

5. Secondary Outcome: Percentage of Participants With Disease Control Rate
Description: Defined as percentage of participants whose best response was PR, CR, or SD as determined by the investigator. SD=Neither PR or PD are met, taking the smallest sum of the LD recorded at baseline as reference. Refer to outcome measure 1 for definition of CR or PR and refer to outcome measure 4 for definition of PD. A 2-sided 95% CI was computed using Clopper-Pearson method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
percentage of participants | 65.4 [50.9 to 78.0]

6. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs), and AEs Leading to Discontinuation of Study Therapy Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0
Description: AE: New untoward medical occurrence or worsening of a preexisting medical condition that does not have causal relationship with this treatment. SAE: Untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, drug dependency/abuse; life-threatening, an important medical event, a congenital anomaly/birth defect; requires inpatient hospitalization/prolongs existing hospitalization. Grade (GR) 3=Severe; and GR4=Life-threatening or disabling. DR=Drug-related. Any Peripheral Neuropathy includes peripheral sensory and motor neuropathies, including muscle weakness, and hypoaesthesia.
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug. Median time on ixapebilone therapy was 10.5 weeks (range: 3 to 30 weeks)
Population: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
participants
  Death (due to disease progression) | 16
  Death (due to pneumonia) | 1
  Death within 30 days of last dose of study therapy | 4
  At least one SAE (Any GR) | 30
  At least one SAE (GR 3-4) | 21
  At least one DR SAE (Any GR) | 12
  At least one DR SAE (GR 3-4) | 9
  At least one AE (Any GR) | 52
  At least one AE (GR 3-4) | 41
  At least one DR AE (Any GR) | 50
  At least one DR AE (GR 3-4) | 31
  AEs leading to study drug discontinuation (Any GR) | 10
  AEs leading to study drug discontinuation (GR 3-4) | 7
  DRAEs leading to study drug discontinuation:Any GR | 4
  DRAEs leading to study drug discontinuation: GR3-4 | 4
  Any Peripheral Neuropathy (Any GR) | 33
  Any Peripheral Neuropathy (GR 3-4) | 4
  DR Peripheral Neuropathy (Any GR) | 32
  DR Peripheral Neuropathy (GR 3-4) | 4

7. Other Pre Specified Outcome: Number of Participants With Best Response as Assessed With Modified RECIST
Description: Best overall response that any participant can have is the best response recorded from the start of treatment until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference). PR: At least 30% reduction from baseline in the sum of the LD of all target lesions. PR criteria should be met again after 4 weeks and before 6 weeks. Stable disease (SD)=Neither PR or progressive disease (PD) are met, taking the smallest sum of the LD recorded at baseline as reference. Refer to outcome measure 4 for definition of PD.
Time Frame: During treatment, assessed every 6 weeks (± 1 week) starting from the 1st dose of therapy until disease progression, or development of intolerable toxicity, for a maximum of 8 cycles (to a maximum follow up for tumor response of 30 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
participants
  Partial Response | 8
  Stable Disease | 26
  Progressive Disease | 15
  Unable to Determine (No tumor assessment) | 1
  Unable to Determine (Other) | 2

8. Secondary Outcome: Number of Participants With Hematology Abnormalities
Description: Grading: NCI CTCAE, Version 3.0. GR1=mild, GR2=moderate, GR3=severe, GR4=life threatening or disabling. Normal ranges provided by local laboratory and may also vary by age and sex. White blood cell (WBC):GR1=<LLN-3.0*10^9/L; GR2=<3.0-2.0*10^9/L; GR3=<2.0-1.0*10^9/L; GR4=<1.0*10^9/L. Absolute Neutrophil Count (ANC):GR1=<LLN-1.5*10^9 /L; GR2=<1.5-1.0*10^9/L; GR3=<1.0-0.5*10^9/L; GR4=<0.5*10^9/L. Platelets:GR1=<LLN-75.0*10^9/L; GR2=<75.0-50.0*10^9/L; GR3=<50.0-25.0*10^9/L, GR4=<25.0*10^9/L. Hemoglobin:GR1=<LLN-10.0g/dL; GR2=<10.0-8.0g/dL; GR3=<8.0-6.5g/dL, GR4=<6.5g/dL. LLN=lower limit of normal.
Time Frame: Assessed once every week for first 3 weeks, as clinically indicated, start of each 3 week cycle (maximum time that any participant was on therapy was 30 weeks).
Population: Participants who received at least 1 dose of ixabepilone and had at least one measurement available during the study therapy period.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
participants
  WBC GR1 | 6
  WBC GR2 | 17
  WBC GR3 | 20
  WBC GR4 | 5
  ANC GR1 | 4
  ANC GR2 | 7
  ANC GR3 | 16
  ANC GR4 | 21
  Platelet Count GR1 | 18
  Platelet Count GR2 | 3
  Platelet Count GR3 | 4
  Platelet Count GR4 | 0
  Hemoglobin GR1 | 17
  Hemoglobin GR2 | 23
  Hemoglobin GR3 | 11
  Hemoglobin GR4 | 0

9. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities
Description: Grading: NCI CTCAE, Version 3.0. GR1=mild, GR2=moderate, GR3=severe, GR4=life threatening or disabling. Normal ranges provided by local laboratory and may also vary by age and sex. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST): GR1=>ULN-2.5*ULN; GR2=>2.5-5.0*ULN; GR3=>5.0-20.0*ULN; GR4=>20.0*ULN. Total bilirubin: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3-10*ULN, GR4=>10*ULN. Creatinine: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3.0-6.0*ULN, GR4=>6.0*ULN. ULN=upper limit of normal.
Time Frame: Assessed within 2 weeks of first dose and every 3 weeks before therapy dose (maximum time that any participant was on therapy was 30 weeks).
Population: Participants who received at least 1 dose of ixabepilone. n=number of participants with at least 1 measurement available during the study therapy period.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 IV
Number analyzed (Participants) | 52
participants
  ALP GR1 (n=49) | 22
  ALP GR2 (n=49) | 1
  ALP GR3 (n=49) | 1
  ALP GR4 (n=49) | 1
  AST GR1 (n=49) | 9
  AST GR2 (n=49) | 0
  AST GR3 (n=49) | 0
  AST GR4 (n=49) | 0
  ALT GR1 (n=50) | 8
  ALT GR2 (n=50) | 1
  ALT GR3 (n=50) | 0
  ALT GR4 (n=50) | 0
  Total bilirubin GR1 (n=49) | 0
  Total bilirubin GR2 (n=49) | 3
  Total bilirubin GR3 (n=49) | 0
  Total bilirubin GR4 (n=49) | 0
  Creatinine GR1 (n=51) | 4
  Creatinine GR2 (n=51) | 1
  Creatinine GR3 (n=51) | 0
  Creatinine GR4 (n=51) | 0

ADVERSE EVENTS:
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug. Median time on ixapebilone therapy was 10.5 weeks (range: 3-30 weeks)
Arm/Group | Ixabepilone 40 mg/m^2 IV
Serious Adverse Events (participants affected / at risk) | 30/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 40 mg/m^2 IV (N=52)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
ANAL ABSCESS (Infections and infestations) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 3
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 6
MUCOSAL INFLAMMATION (General disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
HYPOPHAGIA (Metabolism and nutrition disorders) | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1
PNEUMONIA (Infections and infestations) | 2
PYREXIA (General disorders) | 3
ILEUS (Gastrointestinal disorders) | 2
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2
MALABSORPTION (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 40 mg/m^2 IV (N=52)
HAEMOGLOBIN DECREASED (Investigations) | 4
HYPOAESTHESIA (Nervous system disorders) | 6
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 26
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11
CHEST PAIN (General disorders) | 3
DIARRHOEA (Gastrointestinal disorders) | 20
HEADACHE (Nervous system disorders) | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 25
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 33
MUCOSAL INFLAMMATION (General disorders) | 3
NAUSEA (Gastrointestinal disorders) | 15
ANAEMIA (Blood and lymphatic system disorders) | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7
DYSGEUSIA (Nervous system disorders) | 6
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 6
PYREXIA (General disorders) | 8
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3
CONSTIPATION (Gastrointestinal disorders) | 14
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 9
WEIGHT DECREASED (Investigations) | 11
DIZZINESS (Nervous system disorders) | 8
FATIGUE (General disorders) | 24
LYMPHOPENIA (Blood and lymphatic system disorders) | 3
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 35
INSOMNIA (Psychiatric disorders) | 8
VOMITING (Gastrointestinal disorders) | 10
ABDOMINAL PAIN (Gastrointestinal disorders) | 10
ASTHENIA (General disorders) | 7
LEUKOPENIA (Blood and lymphatic system disorders) | 12
MYALGIA (Musculoskeletal and connective tissue disorders) | 12
RASH (Skin and subcutaneous tissue disorders) | 19
STOMATITIS (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.